CLINICAL TRIAL: NCT00060840
Title: The Effects of Nitric Oxide for Inhalation During Left Ventricular Assist Device (LVAD) Implantation
Brief Title: The Effects of Nitric Oxide for Inhalation During Left Ventricular Assists Device (LVAD) Implantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INOT 41
Record Dates: First submitted 2003-05-14; First posted 2003-05-15 (Estimated); Results first posted 2010-09-17 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Congestive Heart Failure
Keywords: Left Ventricular Assist Device Implantation; Progressive Left Ventricular Failure
MeSH Terms: conditions — Heart Failure | interventions — Nitric Oxide; Endothelium-Dependent Relaxing Factors; Nitrogen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Nitric Oxide (Active Comparator): Inhaled Nitric Oxide (iNO) at 40 parts per million (ppm)
  Interventions: Drug: Nitric Oxide
- Nitrogen (Placebo Comparator): Nitrogen (N2) administered at 40 ppm.
  Interventions: Drug: Nitrogen

INTERVENTIONS:
Drug: Nitric Oxide — 40 ppm of Nitric Oxide continuously administered for 48 hours
  Other Names: INOmax
  Arms: Inhaled Nitric Oxide
Drug: Nitrogen — Nitrogen (N2) administered at 40 ppm for 48 hours
  Arms: Nitrogen

SUMMARY:
The purpose of this study is to assess the utility of nitric oxide for inhalation during left ventricular assist device (LVAD) implantation following cardiopulmonary bypass (CPB). This is to be assessed by the number of patients in each treatment group meeting failure criteria within 24 hours on study drug, as defined by two or more of the following:

* Left ventricular flow rate index (LVFRI) ≤ 2.0 L/min/m^2
* Administration of ≥ 20 inotropic equivalents (IE)

  * 10 µg/kg/min dopamine, dobutamine, enoximone or amrinone is equivalent to 10 IE
  * 0.1 µg/kg/min epinephrine or norepinephrine is equivalent to 10 IE
  * 1 µg/kg/min milrinone is equivalent to 15 IE
  * 0.1 U/min vasopressin is equivalent to 10 IE
* Mean arterial pressure (MAP) ≤ 55 mmHg
* Central venous pressure (CVP) ≥ 16 mmHg
* Percent mixed venous oxygen saturation (SvO2) ≤ 55%

Or at least one of the following criteria:

* Failure to wean from cardiopulmonary bypass at least once due to hemodynamic failure. Re-initiation of cardiopulmonary bypass to correct bleeding or other technical issues will not be considere 'failure to wean'
* Death

DETAILED DESCRIPTION:
40 ppm of either nitric oxide for inhalation or N2 (placebo) will be continuously administered to the patient starting at least 5 minutes prior to initiating the first weaning attempt from CPB and continue until the patient is either extubated, has reached failure criteria, or has been treated with study drug for 48 hours following discontinuation of CPB, whichever come first.

All patients will be monitored peri-operatively with a pulmonary arterial line, central venous line, and systemic arterial line. Baseline data collection by a designated clinical staff member will begin following induction of anesthesia and prior to skin incision. Following a successful wean from cardiopulmonary bypass, post-op data will be collected within 1 hour following end time of surgery. Data will then be collected at 6, 12, 18, 24, and 48 hours from post-op or until extubation, in which case weaning from study drug will begin.

Open label investigational nitric oxide for inhalation may be administered once a patient meets a minimum of two of the failure criteria or fails to wean at least once due to hemodynamic failure from cardiopulmonary bypass.

ELIGIBILITY:
Inclusion criteria:

* Scheduled to undergo their first LVAD implantation, (or at least 6 months after explanation of a previous LVAD).
* Has a pulmonary vascular resistance of at least 2.5 Wood units (200 dynes/sec.) in the 30 days prior to LVAD placement.
* Greater than 18 years of age.
* Signed IRB approved informed consent.

Exclusion criteria:

* Patients with congestive heart failure due to giant cell myocarditis or restrictive cardiomyopathy.
* Elective Biventricular Assist Device (BiVAD) surgery, or current support with a temporary BiVad.
* LVAD procedure expected to be done without cardiopulmonary bypass.
* Pregnancy (a negative pregnancy test must be documented prior to enrollment).
* Received nitric oxide by inhalation therapy within the past 24 hours.
* Investigational drugs that are expected to change systemic or pulmonary vascular resistance are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-07; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Baldassarre, MD, Study Director — Mallinckrodt
Locations (11):
- United States (8):
  - Newark Beth Isreal Medical Center, Newark, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas/St. Paul Medical Center, Dallas, Texas
  - Texas Heart Institute, Houston, Texas
- Germany (2):
  - Herz-und Diabeteszentrum Nordrhein-Westfalen, Gergstrab, Bad Oeynhausen
  - Deutsches Herfzzentrum Berlin, Augustenburger Platz, State of Berlin
- Harefield Hospital, Harefield, Middlesex, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 8 study medical centers that participated and enrolled subjects; 6 centers in the United States and 2 centers in Germany. There were 150 subjects enrolled in the study.
Groups:
- Inhaled Nitric Oxide: Inhaled Nitric Oxide (iNO) administered through the INOvent delivery system to subjects at 40 parts per million (ppm) for up to 48 hours
- Nitrogen: Nitrogen (N2) administered through the INOvent delivery system to subjects at 40 ppm for up to 48 hours.
Period: Overall Study
Arm/Group | Inhaled Nitric Oxide | Nitrogen
Started | 73 | 77
Completed | 69 | 68
Not Completed | 4 | 9
Not completed — Change in surgical plan | 2 | 6
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Subinvestigator unavailable | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide | Nitrogen | Total
Number analyzed (Participants) | 73 | 77 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 73 | 77 | 150
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (9.75) | 54.0 (11.95) | 55.8 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 64 | 65 | 129
Region of Enrollment [Number; unit: participants]
  United States | 38 | 42 | 80
  Germany | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With Left Ventricular Failure During Left Ventricular Assistance Device (LVAD) Placement After Cardio Pulmonary Bypass, as Determined by Failure Criteria, After Administration of Nitric Oxide.
Description: Failure criteria used to measure outcome includes:
  * Left ventricular flow rate index (LVFRI) ≤ 2.0 L/min/m^2
  * Administration of ≥ 20 inotropic equivalents (IE)
  * Mean arterial pressure (MAP) ≤ 55 mm Hg
  * Central venous pressure (CVP) ≥ 16 mm Hg
  * Percentage of mixed venous oxygen saturation (SvO2) of ≤ 55% OR failure to wean from cardio pulmonary bypass (CPB) at least once due to hemodynamic failure or death.
Time Frame: 28 days
Population: The analysis was determined for intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Inhaled Nitric Oxide | Nitrogen
Number analyzed (Participants) | 73 | 77
Participants | 7 | 12

ADVERSE EVENTS:
Arm/Group | Inhaled Nitric Oxide | Nitrogen
Serious Adverse Events (participants affected / at risk) | 7/73 | 11/77
Other Adverse Events (participants affected / at risk) | 14/73 | 6/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (N=73) | Nitrogen (N=77)
Right Ventricular Failure (Cardiac disorders) | 3 (3) | 3 (3)
Postprocedural hemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Hemorrhage (Vascular disorders) | 1 (1) | 3 (3)
Haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Procedural Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (N=73) | Nitrogen (N=77)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Right Ventricular Dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Central Venous Pressure Decreased (Investigations) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Aspartate Aminotransferase Abnormal (Investigations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Pharyngeal Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemodynamic Instability (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other